CLINICAL TRIAL: NCT05846607
Title: A Deep Learning Approach to Identify Patients With Full Stomach on Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, le tian wang, Doctor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-491
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Gastic Antrum
Keywords: Deep learning，gastric antrum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment (Experimental): The data will be collected in two phases. Firstly, after a fasting period of eight hours, the participants received ultrasound scan by expert doctor with the objective of measuring the fasting gastric antrum area in supine and right lateral decubitus(RLD)position(phase 1).Then the expert made the grading according to the ultrasound image.
  In phase 2, the participant will ingest 0 to 400ml of the study drink described below randomly. The individual will be immediately positioned in the supine position and another ultrasound scan will be carried out. Again in the RLD position.
  Interventions: Dietary Supplement: Intervention oral supplement

INTERVENTIONS:
Dietary Supplement: Intervention oral supplement — The oral supplement used as intervention for the study will be DongzheSutang(DAISY FSMP,Jiangsu,China). The formula contains only carbohydrate:12.5g in 100ml of product(glucose syrup and maltodextrin)，with a caloric density of 16.32kcal/g.

SUMMARY:
Preoperative gastric ultrasonography is a newly developed tool used to evaluate gastric content and volume in assessing perioperative aspiration risk and guide anaesthetic management. And then build up effective clinical predictive models for identification of full stomach, which can predict the high aspiration risk.

DETAILED DESCRIPTION:
Aspiration of gastric contents can be a serious anesthetic related complication. Preoperative fasting was a common practice to decrease perioperative aspiration risk. However，one of most important prescription of enhanced recovery after surgery protocols is the reduction of preoperative fasting time in opposition to the traditional recommendation of overnight fast. Gastric antral sonography prior to anesthesia may have a role in identifying patients at risk of aspiration. The aim of this study is to construct models using deep learning for identification of full stomach, which can predict the aspiration risk.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing surgery Age: 18~85 yeas ASA 1~3

Exclusion Criteria:

-Diabetes mellitus Upper gastrointestinal pathology such as hiatus hernia, oesophageal cancer Prior surgery to upper GI On medication that may affect gastric emptying time Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the model | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Le tian Wang, MD, Principal Investigator — Fudan University affiliated Huashan Hospital
Locations (1):
- Fudan University affiliated Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No